CLINICAL TRIAL: NCT05022901
Title: An Open-Label Expanded Access Study of the Melphalan/Hepatic Delivery System (HDS) in Patients With Hepatic Dominant Ocular Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHP-OCM-501
Record Dates: First submitted 2021-08-18; First posted 2021-08-26 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Ocular Melanoma; Metastatic Uveal Melanoma
Keywords: percutaneous hepatic perfusion; PHP; uveal melanoma; HEPZATO
MeSH Terms: conditions — Uveal Melanoma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Melphalan/HDS (Experimental): Eligible patients will be treated with Melphalan/HDS 3.0 mg/kg Ideal Body Weight (IBW). Melphalan/HDS treatment will be administered every 6 weeks for a total of 6 cycles with an acceptable delay of another 2 weeks before the next planned treatment to allow for recovery of melphalan-related toxicity, if needed.
  Interventions: Combination Product: Melphalan (3 mg/kg IBW) with Hepatic Delivery System (HDS)

INTERVENTIONS:
Combination Product: Melphalan (3 mg/kg IBW) with Hepatic Delivery System (HDS) — Melphalan administered directly to the liver via the Hepatic Delivery System (HDS) infused over a 30 minute period, followed by a 30 minute washout period
  Other Names: percutaneous hepatic perfusion; PHP; HEPZATO

SUMMARY:
Patients in the study will be treated with Melphalan/HDS and will receive up to 6 total treatments.

This study will evaluate the safety and effects of the treatment.

DETAILED DESCRIPTION:
The study will consist of 3 phases:

Screening/Baseline Phase: Screening assessments will be conducted within 28 days prior to the eligibility date to determine each patient's overall eligibility and baseline characteristics. These assessments will include medical history, physical examination, Eastern Cooperative Oncology Group (ECOG) performance status (PS), Quality of Life questionnaire, 12 lead electrocardiogram (ECG), echocardiogram (ECHO), vital signs, full hematology and biochemistry, Quality of Life questionnaire, radiologic assessments of baseline disease status and concomitant medications.

For patients with a history of liver surgery or major vasculature surgery, an angiogram evaluation of their vasculature will be performed for compatibility for Percutaneous Hepatic Perfusion (PHP) prior to confirming eligibility.

Eligibility date: This is the date on which all screening assessments have been completed and the patient is determined to be eligible for the trial.

Treatment Phase: The first study treatment should occur within 14 days of the eligibility date. Eligible patients will be treated with Melphalan/HDS 3.0 mg/kg Ideal Body Weight (IBW). Melphalan/HDS treatment will be administered every 6 weeks for a total of 6 cycles with an acceptable delay of another 2 weeks before the next planned treatment to allow for recovery of melphalan-related toxicity, if needed. Tumor response will be assessed every 12 weeks (+ 2 weeks) until disease progression. Patients with progressive disease (PD) will be discontinued from study treatment, and will continue to be followed until death. Melphalan/HDS treatment will also be discontinued if recovery from treatment related toxicity requires more than 8 weeks from the last treatment. An end-of-treatment visit (EOT) will be conducted approximately 6 to 8 weeks following the final study treatment.

Follow-up Phase: Once the patient has completed the end-of-treatment (EOT) visit in accordance with the schedule of events they will enter the follow-up phase. If the disease has not progressed at the EOT, the patient will need to continue with disease assessment visits every 12 weeks (± 2 weeks) until disease progression is documented. After disease progression, follow-up is to be by phone every 3 months for survival status until death.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Patients must weigh ≥ 35 kg (due to possible size limitations with respect to percutaneous catheterization of the femoral artery and vein using the Delcath Hepatic Delivery System).
3. 50% or less histologically or cytologically-proven ocular melanoma metastases in the parenchyma of the liver.
4. Disease in the liver must be measurable by computed tomography (CT) and/or magnetic resonance imaging (MRI).
5. Evidence of limited extrahepatic disease on preoperative radiological studies is acceptable if the life-threatening component of disease is in the liver. Limited extrahepatic disease is defined in this protocol as follows: metastasis in bone, subcutaneous, lung or lymph nodes that is amenable to resection or radiation and has a defined treatment plan. Patients with extra-hepatic tumor burden which does not have a defined treatment plan (i.e. monitor or is unable to be resected or radiated) must not be included in the trial.
6. Scans used to determine eligibility (CT scan of the chest/abdomen/pelvis and MRI of the liver) must be performed within 28 days prior to eligibility. An MRI of the liver is required at screening to validate that CT accurately reflects the extent of disease in the liver. For patients with MRI intolerance, a 3-phase liver CT is to be done in place of liver MRI.
7. Patients must not have had chemotherapy, radiotherapy, chemoembolization, radioembolization, or immunoembolization for their malignancy within 30 days prior to treatment and must have recovered from all side effects of therapeutic and diagnostic interventions except those listed in Appendix B of the study protocol.
8. Patients receiving anti programmed cell death protein 1 (PD-1) immunotherapy such as pembrolizumab or nivolumab, or human cytotoxic T-lymphocyte antigen 4 blocking antibody such as ipilimumab must have completed treatment 8 weeks prior to study eligibility.
9. Patients must have an ECOG PS of 0-1 at screening.
10. Patients must have adequate hepatic function as evidenced by total serum bilirubin ≤1.5 x the upper limit of normal (ULN) and a prothrombin time (PT) within 2 seconds of the upper normal limit. Aspartate aminotransferase/alanine aminotransferase (AST/ALT) must be ≤ 2.5 x ULN.
11. Patients must have a platelet count > 100,000/µL, hemoglobin ≥ 10.0 gm/dL, white blood cell count (WBC) > 2,000/uL, absolute neutrophil count ≥ 1.5 x 109/L, and a serum creatinine ≤ 1.5 mg/dL unless the measured creatinine clearance is > 40 mL/min/1.73 m2.
12. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (β-human chorionic gonadotropin) within 7 days prior to eligibility.
13. Provided signed informed consent.

Exclusion Criteria:

1. Patients with Child-Pugh Class B or C cirrhosis or with evidence of portal hypertension by history, endoscopy, or radiologic studies.
2. Those with New York Heart Association functional classification II, III or IV active cardiac conditions, including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), worsening or new-onset congestive heart failure, significant arrhythmias and severe valvular disease must be evaluated for risks of undergoing general anesthesia.
3. History or evidence of clinically significant pulmonary disease that precludes the use of general anesthesia.
4. Women of childbearing potential (WOCBP) i.e. fertile meaning not permanently sterilized and having had a menstrual period within the past 12 months) unable to undergo hormonal suppression to avoid menstruation during treatment.
5. WOCBP and fertile males (not permanently sterile by bilateral orchiectomy) unwilling or unable to use highly effective contraception method from consent to at least 6 months after the last administration of study treatment (e.g. combined hormonal contraception; progestogen-only hormonal contraception; Intrauterine device, intrauterine hormone-releasing system; bilateral tubal occlusion, vasectomized partner or sexual abstinence).
6. Females that are pregnant or are breastfeeding.
7. Patients taking immunosuppressive drugs; however, oral corticosteroids ≤ 10 mg/ day are allowed.
8. Patients who are unable to be temporarily removed from chronic anti-coagulation therapy.
9. Patients with active bacterial infections with systemic manifestations (malaise, fever, leucocytosis) are not eligible until completion of appropriate therapy.
10. Patients with severe allergic reaction to iodine contrast, which cannot be controlled by premedication with antihistamines and steroids.
11. Patients with a history of or known hypersensitivity to melphalan or the components of the Melphalan/HDS system.
12. Patients with latex allergy.
13. Patients with a history of hypersensitivity to heparin or the presence of heparin-induced thrombocytopenia.
14. Patients with a history of bleeding disorders or evidence of intracranial abnormalities which would put them at risk for bleeding with anti-coagulation (e.g., strokes, active metastases).
15. Patients with a history of gastrinoma, NOTE: For patients with a history of liver surgery or major vasculature surgery, a CT angiogram or MR angiogram is required during screening to assure the patient does not have hepatic vasculature incompatible with perfusion, hepatofugal flow in the portal vein or known unresolved venous shunting.
16. Known varices at risk of bleeding, including medium or large esophageal or gastric varices, or active peptic ulcer.
17. Patients with prior Whipple's procedure.
18. Patients with brain metastases or presence of other intracranial lesions at risk for bleeding by history or baseline radiologic imaging.
19. Patients with an active infection, including Hepatitis B and Hepatitis C infection. Patients with anti-hepatitis B core antibody (HBc) positive, or hepatitis B surface antigen (HBsAg) but DNA negative are exception(s).
20. Uncontrolled endocrine disorders including diabetes mellitus, hypothyroidism, or hyperthyroidism.
21. Received any investigational agent for any indication within 30 days prior to first treatment.
22. Not recovered from side effects of prior therapy to ≤ Grade 1 (according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v. 5.0). Certain side effects that are unlikely to develop into serious or life-threatening events (e.g. alopecia) are allowed at > Grade 1.
23. Cancers other than ocular melanoma for which the patient is currently under treatment or still deemed to be not cancer free.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From eligibility until death due to any cause, for up to 104 weeks
  The number and type of adverse events will be assessed per CTCAE version 5.0.

SECONDARY OUTCOMES:
Efficacy (ORR) | Every 12 (+/-2) weeks until progression, for up to 104 weeks
  Defined as the proportion of patients with a best overall response (BOR) based on a confirmed complete response or partial response (CR+PR) determined by the investigator per the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Efficacy (OS) | From eligibility until death due to any cause, for up to 104 weeks
  The time from the eligibility date to date of death due to any cause
Efficacy (PFS) | Every 12 (+/-2) weeks until progression, for up to 104 weeks
  The time from the eligibility date to the first documented progression or death due to any cause determined by the investigator
Quality of Life (FHSI-8) | Every 6-8 weeks until the end of treatment, for up to 52 weeks
  FHSI-8 Quality of Life Survey

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford Cancer Institute, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Tennessee Health Science Center, Memphis, Tennessee